CLINICAL TRIAL: NCT02889952
Title: Parathyroid Autofluorescence Visualization During Thyroid Surgery: Impact on Postoperative Hypocalcemia
Brief Title: Clinical Impact of Parathyroid Autofluorescence Visualization During Thyroid Surgery
Status: Completed | Type: Observational
Sponsor: Hôpital Européen Marseille (Other)
Collaborators: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Principal Investigator, Fares BENMILOUD, Dr, Hôpital Européen Marseille
Other Study IDs: ParaFluo1
Record Dates: First submitted 2016-08-29; First posted 2016-09-07 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-08

CONDITIONS: Hypocalcemia
Keywords: postoperative hypocalcemia; near infrared imaging; parathyroid autofluorescence
MeSH Terms: conditions — Hypocalcemia

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- NIR-: All consecutive patients (n=174) who underwent conventional total thyroidectomy (TT)+/- lymph node dissection (LND) without the use of NIR - parathyroid identification was done by naked eye only- by surgeon 1, from January 2015 to January 2016 (period 1)
- NIR: All consecutive patients (n=63) who underwent conventional total thyroidectomy (TT)+/- lymph node dissection (LND) with intraoperative use of NIR - surgical field was examined with NIR before any thyroid dissection- by surgeon 1, from February 2016 to May 2016 (period 2)
  Interventions: Device: Near infrared camera (NIR)
- Control1: Patients (n=30) patients randomly selected among the patients who underwent TT+/- LND without the use of NIR, by another surgeon in the unit (surgeon 2), during period 1.
- Control2: Patients (n=30) patients randomly selected among the patients who underwent TT+/- LND without the use of NIR, by surgeon 2, during period 2.

INTERVENTIONS:
Device: Near infrared camera (NIR) — Surgical field was examined with NIR, during a few minutes (<5') with room lights switched off, to avoid parasite lights, then conventional open thyroidectomy was resumed conventionally. Real-time images, evocative of autofluorescent parathyroids, were checked visually.
  NIR consisted of a 750 nm class 1 laser excitation, with a power <20mW/cm2 (5 times less than the limit of 100mw/cm2, fixed by the international norm IEC 60601-2-41). It was provided by the Fluobeam® camera, which was inserted into a sterile cover and hold at a 15-20 cm distance from the patient. The system has an FDA 510(k) authorization for clinical use in parathyroid surgery and a European Community certification (Class 1 device).
  Other Names: Fluobeam® system (Fluoptics®, Grenoble, France)
  Groups: NIR

SUMMARY:
This Before-and-after Controlled Study study evaluates the clinical impact of parathyroid autofluorescence visualization using near infrared light (NIR) during total thyroidectomy (TT).

It compares two groups of consecutive patients who underwent TT associated or not to lymph node dissection (LND) with and without intraoperative use of NIR, by the same surgeon.

DETAILED DESCRIPTION:
Total thyroidectomy (TT) is responsible for postoperative hypocalcemia in 20-30% of patients, which is definitive in 1-4% of operated patients (1).

This complication is mainly due to surgery-induced parathyroid dysfunction, which could be improved by a better intraoperative identification of the parathyroids.

Intraoperative parathyroid auto-fluorescence visualization (without any dye injection) using near infrared light (NIR) is an emerging technique, which allows correct identification of normal parathyroids in almost all cases (2), but the clinical impact of NIR is unknown.

The main objective of this study is to assess the impact of intraoperative use of NIR camera on postoperative hypocalcemia. Secondary objectives are to assess the impact of NIR on the visualization, autotransplantation and inadvertent resection rates during TT.

The investigators compare 2 groups of patients operated by one surgeon during 2 consecutive but distinct periods (before and after the use of NIR) with control groups operated by another surgeon during the same periods. This study is observational since there was no predefined protocol nor sample size calculation of study groups prior to data collection.

ELIGIBILITY:
Inclusion Criteria:

* All patients who underwent one-stage total thyroidectomy, associated or not to lymph node dissection (TT +/- LND)

Exclusion Criteria:

* Combined parathyroid and thyroid disease (including patients with enlarged parathyroids incidentally found during surgery and resected)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who underwent one-stage total thyroidectomy, associated or not to lymph node dissection (TT +/- LND) in the European Hospital Marseilles were consecutively included in this study, from January 2015 to May 2016.
Sampling Method: Probability Sample
Enrollment: 297 (Actual)
Dates: Start 2015-01; Primary Completion 2016-05 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Postoperative hypocalcemia | 6 months
  Postoperative day 1 and day 2 corrected calcemia(hypocalcemia when calcemia <2mmol/l). If hypocalcemia, calcium is measured at 1 month and 6 months

SECONDARY OUTCOMES:
number of identified parathyroids | immediate (intraoperative)
number of autotransplantated parathyroids | immediate (intraoperative)
  when parathyroids are impossible to preserve in situ, they are fragmented and inserted in the sternocleidomastoid muscle
number of inadvertently resected parathyroids | within 15 days after surgery (time to complete pathology examination)
  When parathyroids are found on the thyroid specimen during pathology examination, they are called 'inadvertently resected'

OTHER OUTCOMES:
number of parathyroids identified by NIR before naked eye | immediate (intraoperative)
  in NIR group only

CONTACTS AND LOCATIONS:
Overall Officials: Fares BENMILOUD, MD, Principal Investigator — Hopital Europeen Marseille

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Duclos A, Peix JL, Colin C, Kraimps JL, Menegaux F, Pattou F, Sebag F, Touzet S, Bourdy S, Voirin N, Lifante JC; CATHY Study Group. Influence of experience on performance of individual surgeons in thyroid surgery: prospective cross sectional multicentre study. BMJ. 2012 Jan 10;344:d8041. doi: 10.1136/bmj.d8041. PMID 22236412
- [Background] McWade MA, Sanders ME, Broome JT, Solorzano CC, Mahadevan-Jansen A. Establishing the clinical utility of autofluorescence spectroscopy for parathyroid detection. Surgery. 2016 Jan;159(1):193-202. doi: 10.1016/j.surg.2015.06.047. Epub 2015 Oct 9. PMID 26454675